CLINICAL TRIAL: NCT02800304
Title: More-2-Eat; Implementation of INPAC
Acronym: m2E
Status: Completed | Type: Observational
Sponsor: University of Waterloo (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Heather Keller, Research Chair, Nutrition & Aging, University of Waterloo
Other Study IDs: 20590
Record Dates: First submitted 2016-06-07; First posted 2016-06-15 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Acute Care Medical
Keywords: malnutrition; food intake; frailty
MeSH Terms: conditions — Malnutrition; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
M2E is a developmental evaluation of the implementation of the Integrated Nutrition Pathway for Acute Care, in five medical units in five hospitals in Canada.

ELIGIBILITY:
Inclusion Criteria:

* admitted to study unit
* no delirium or dementia
* return to community anticipated

Exclusion Criteria:

* unable to communicate in English or French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: medical patients over the age of 18 years
Sampling Method: Non-Probability Sample
Enrollment: 5995 (Actual)
Dates: Start 2015-09-01; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Implementation success of Integrated Nutrition Pathway for Acute Care (INPAC) | admission
  INPAC is an evidence based pathway to improve detection, prevention and treatment of malnutrition in acute care. The primary outcome of this study is the trajectory and proportion of care activities that happen for a given population e.g. % screened, assessed with SGA, have standard care strategies provided etc.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Keller, PhD, Principal Investigator — University of Waterloo
Locations (5):
- Canada (5):
  - Royal Alexander Hospital, Edmonton, Alberta
  - Concordia Hospital, Winnipeg, Manitoba
  - Niagara Health Systems, Niagara Falls, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Pasqua Hospital, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laur C, Bell J, Valaitis R, Ray S, Keller H. The role of trained champions in sustaining and spreading nutrition care improvements in hospital: qualitative interviews following an implementation study. BMJ Nutr Prev Health. 2021 Sep 28;4(2):435-446. doi: 10.1136/bmjnph-2021-000281. eCollection 2021. PMID 35028514
- [Derived] Valaitis R, Laur C, Keller H, Butterworth D, Hotson B. Need for the Integrated Nutrition Pathway for Acute Care (INPAC): gaps in current nutrition care in five Canadian hospitals. BMC Nutr. 2017 Jul 14;3:60. doi: 10.1186/s40795-017-0177-8. eCollection 2017. PMID 32153840
- [Derived] Laur C, Bell J, Valaitis R, Ray S, Keller H. The Sustain and Spread Framework: strategies for sustaining and spreading nutrition care improvements in acute care based on thematic analysis from the More-2-Eat study. BMC Health Serv Res. 2018 Dec 4;18(1):930. doi: 10.1186/s12913-018-3748-8. PMID 30509262
- [Derived] Keller HH, Xu Y, Dubin JA, Curtis L, Laur CV, Bell J; More-2-Eat Team. Improving the standard of nutrition care in hospital: Mealtime barriers reduced with implementation of the Integrated Nutrition Pathway for Acute Care. Clin Nutr ESPEN. 2018 Dec;28:74-79. doi: 10.1016/j.clnesp.2018.09.075. Epub 2018 Oct 11. PMID 30390896
- [Derived] Keller HH, Valaitis R, Laur CV, McNicholl T, Xu Y, Dubin JA, Curtis L, Obiorah S, Ray S, Bernier P, Gramlich L, Stickles-White M, Laporte M, Bell J. Multi-site implementation of nutrition screening and diagnosis in medical care units: Success of the More-2-Eat project. Clin Nutr. 2019 Apr;38(2):897-905. doi: 10.1016/j.clnu.2018.02.009. Epub 2018 Mar 22. PMID 29605573
- [Derived] Laur C, Valaitis R, Bell J, Keller H. Changing nutrition care practices in hospital: a thematic analysis of hospital staff perspectives. BMC Health Serv Res. 2017 Jul 19;17(1):498. doi: 10.1186/s12913-017-2409-7. PMID 28724373
- See also: Primary analysis on implementation process — http://doi.org/10.1016/j.clnu.2018.02.009
- See also: Primary analysis on patient outcomes resulting from implementation — http://doi.org/10.1016/j.clnesp.2018.09.075

DOCUMENTS (1):
  • Study Protocol (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT02800304/Prot_000.pdf